CLINICAL TRIAL: NCT03652441
Title: Consolidation Therapy With Brentuximab Vedotin After Allogeneic Stem Cell Transplantation for Relapsed or Refractory Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Christoph Scheid, Head of Stem Cell Transplantation, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Koeln 3263; 2018-000873-59 (EudraCT Number)
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Classical Hodgkin Lymphoma
MeSH Terms: interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maintenance (Experimental): Brentuximab Vedotin will be administered i.v. at 1.8mg/kg at 3-weekly intervals for up to 16 infusions
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — BV will be administered i.v. at 1.8mg/kg at 3-weekly intervals for up to 16 infusions
  Other Names: BV

SUMMARY:
The aim of the trial is to improve disease control after an allogeneic stem cell transplantation (alloSCT) for relapsed or refractory classical Hodgkin lymphoma (rrHL, cHL) with consolidation therapy by Brentuximab Vedotin (BV) for up to one year.

The primary objective of the trial is to show efficacy of the experimental consolidative treatment strategy. Secondary objectives are to further evaluate efficacy, show safety and feasibility and perform correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory cHL who receive an allogeneic stem cell transplantation
* Histologically proven cHL in the most recent tumor biopsy
* Absolute neutrophil count ≥ 500/mm³
* ECOG ≤2
* Age ≥ 18 years

Exclusion Criteria:

* Presence of nodular lymphocyte-predominant HL (NLPHL) or grey-zone lymphoma
* Progressive disease as last documented response prior to alloSCT
* Any peripheral neuropathy ≥ grade 2
* Any other serious disease or organ dysfunction which might impair protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2019-11-13 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
1-year Cumulative incidence of relapse (CIR) | 1 year
  1-year Cumulative incidence of relapse (CIR)

SECONDARY OUTCOMES:
1- and 2-year Progression-free survival (PFS) | 1 and 2 years
  1- and 2-year Progression-free survival (PFS)

CONTACTS AND LOCATIONS:
Overall Officials: Christof Scheid, Prof., Principal Investigator — University of Cologne, I. Dept. of Medicine
Locations (1):
- 1st Department of Medicine, Cologne University Hospital, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided